CLINICAL TRIAL: NCT05059951
Title: Chemotherapy With or Without Immune Checkpoint Inhibitors for Lung Cancer
Acronym: CREATE
Status: Recruiting | Type: Observational
Sponsor: Hunan Province Tumor Hospital (Other)
Responsible Party: Principal Investigator, Yongchang Zhang, Professor, Director of Clinical Trial Center, Hunan Province Tumor Hospital
Other Study IDs: 20210113
Record Dates: First submitted 2021-09-17; First posted 2021-09-28 (Actual); Last update posted 2024-06-04 (Actual); Status verified 2024-06

CONDITIONS: Non Small Cell Lung Cancer
Keywords: Chemotherapy, Immune Checkpoint Inhibitors
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Immune Checkpoint Inhibitors; Drug Therapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — tissue sample and plasma DNA was obtained with the permission of patients.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (12):
- Cohort A: Extansive Stage Small Cell Lung Cancer treated with first line Chemotherapy with or without Checkpoint Inhibitors .
  Interventions: Drug: Immune checkpoint inhibitor
- Cohort B: Limit Stage Small Celll Lung Cancer treated with first line Chemotherapy with or without Checkpoint Inhibitors .
  Interventions: Drug: Immune checkpoint inhibitor
- Cohort C: Small Celll Lung Cancer who progressed from first line treatment and received subsequential Chemotherapy with or without Checkpoint Inhibitors.
  Interventions: Drug: Immune checkpoint inhibitor
- Cohort D: Metastastic Non-small cell Lung Cancer treated with first line Chemotherapy with or without Checkpoint Inhibitors.
  Interventions: Drug: Immune checkpoint inhibitor
- Cohort E: Metastastic Non-small cell Lung Cancer who progressed from first line treatment and received subsequential Chemotherapy with or without Checkpoint Inhibitors.
  Interventions: Drug: Immune checkpoint inhibitor
- Cohort F: Resectable Non-small cell Lung Cancer treated with first line Chemotherapy with or without Checkpoint Inhibitors.
  Interventions: Drug: Immune checkpoint inhibitor
- Cohort G: Unresectable Non-small cell Lung Cancer treated with first line Chemotherapy with or without Checkpoint Inhibitors.
  Interventions: Drug: Immune checkpoint inhibitor
- Cohort H: Non-small cell Lung Cancer received neoadjuvent or adjuvent Chemotherapy with or without Checkpoint Inhibitors.
  Interventions: Drug: Immune checkpoint inhibitor
- Cohort I: Cohort I, Non-small cell Lung Cancer with EGFR, ALK and ROS1 sensitive mutation who received Chemotherapy with or without Checkpoint Inhibitors.
  Interventions: Drug: Immune checkpoint inhibitor
- Cohort J: Non-small cell Lung Cancer with other oncogenic mutation including RET, BRAF etc who received Chemotherapy with or without Checkpoint Inhibitors.
  Interventions: Drug: Immune checkpoint inhibitor
- Cohort K: Non-small cell Lung Cancer received Chemotherapy plus bevacizumab with or without Checkpoint Inhibitors.
  Interventions: Drug: Immune checkpoint inhibitor
- Cohort L: Non-small cell Lung Cancer who enrolled in clinical trials.
  Interventions: Drug: Immune checkpoint inhibitor

INTERVENTIONS:
Drug: Immune checkpoint inhibitor — Chemotherapy follow the guild line.
  Other Names: Chemotherapy

SUMMARY:
Although several clinical trials provide evidence for efficacy benefit for Checkpoint Inhibitors plus chemotherapy for lung cancer. However, there was rare evidence for clinical evidence in Hunan province.

DETAILED DESCRIPTION:
This prospective study aimed to assess its efficacy and adverse event for Checkpoint Inhibitors with or without chemotherapy in clincial practice. Several cohorts were devided including pathological type, treatment line, treatment regiems, combination strategies. Tissue samples were collected with permission of patients for TME evaluation.

ELIGIBILITY:
Inclusion Criteria:

1. ≥18，Lung Cancer Confirmed by Histopathology
2. Treated with Chemotherapy with or Without Checkpoint Inhibitors.
3. ECOG 0 - 1.
4. Predicted survival ≥ 12 weeks.
5. Adequate bone marrow hematopoiesis and organ function
6. Presence of measurable lesions according to RECIST 1.1.
7. Subjects with stable brain metastases may be included in the study.

Exclusion Criteria:

Patients did not match for the Inclusion Criteria.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Chemotherapy With or Without Immune Checkpoint Inhibitors for Lung Cancer
Sampling Method: Probability Sample
Enrollment: 15000 (Estimated)
Dates: Start 2021-10-03 (Actual); Primary Completion 2026-09-15 (Estimated); Study Completion 2028-03-01 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) | Time from first subject dose to study completion, or up to 36 month
  To assess progression-free survival of patients treated by different treatment according to Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1 by investigator, define as first dose to first documented disease progression assessed by investigator or death due to any cause

SECONDARY OUTCOMES:
Overall survival (OS) | Time from first subject dose to study completion, or up to 36 months.
  To assess overall survival, define as first dose to the death of the subject due to any cause
Objective Response Rate (ORR) | Time from first subject dose to study completion, or up to 36 months.
  To assess ICI and TKIs overall response rate according to Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1
Duration of Response (DOR) | Time from first subject dose to study completion, or up to 36 month
  To assess duration of response for subjects with CR or PR according to Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1 by investigator , defined as the time from the first documented CR or PR to disease progression or death
Adverse events (AEs) according to CTCAE 5.0 | From first dose until 28 days after the last dose, up to 24 month
  Number of participants with adverse events (AEs) according to CTCAE 5.0
Patient reported outcome | Time from first subject dose to study completion, or up to 36 months.
  Patient reported outcomes (PROs): A report that directly reflects a patient's assessment of their own health status.

CONTACTS AND LOCATIONS:
Overall Officials: Yongchang Zhang, MD, Principal Investigator — Hunan Cancer Hospital
Locations (1):
- Hunan Cancer Hospital, Changsha, Hunan, China